CLINICAL TRIAL: NCT06809478
Title: Clinical and Radiographic Evaluation of Chitosan Versus Formocresol After Vital Pulpotomy of Primary Molars: a Randomized Clinical Study
Brief Title: Clinical and Radiographic Evaluation of Chitosan Versus Formocresol After Vital Pulpotomy of Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reem Ibrahim Helmi, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS Pulpotomy
Record Dates: First submitted 2025-01-16; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis - Reversible; Pulpotomy
Keywords: pulpotomy; formocresol; chitosan; primary molars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pulpotomy using Chitosan (Experimental): Chitosan is a natural cationic polysaccharide polymer obtained from chitin deacetylation. It is a linear biopolymer consisting of 2-amino-2-deoxy-β-D-glucose (60-100%) and 2-acetamino -2-deoxy-β-D-glucoside (0-50%) bound together by ß (1→4) bonds. It is biocompatible and has antibacterial, anti-inflammatory and hemostatic properties.
  Interventions: Procedure: Pulpotomy using Chitosan liquid
- Pulpotomy using Formocresol (Active Comparator): Buckley's formocresol is composed of 31% water base, 15% glycerin to prevent formaldehyde from polymerizing to paraformaldehyde, 19% formaldehyde as an alkylating agent, and 35% tricresol as a protein-coagulating phenolic substance. A 1:5 concentration of Buckley's formocresol is used in this trial.
  Interventions: Procedure: Pulpotomy using Formocresol

INTERVENTIONS:
Procedure: Pulpotomy using Chitosan liquid — 1. After complete hemostasis, a cotton pellet damp with chitosan liquid will be applied and gently placed over the pulp stumps for 5 minutes and removed. Then, a thick mix of zinc oxide and eugenol will be placed and gently condensed into the pulp chamber by a moistened cotton pellet.
  2. Tooth will be restored with stainless steel crown.
  Other Names: Chitosan Pulpotomy
  Arms: Pulpotomy using Chitosan
Procedure: Pulpotomy using Formocresol — 1. After complete hemostasis, a cotton pellet damp with formocresol will be applied and gently placed over the pulp stumps for 5 minutes and removed. Then, a thick mix of zinc oxide and eugenol will be placed and gently condensed into the pulp chamber by a moistened cotton pellet.
  2. Tooth will be restored with stainless steel crown.
  Other Names: Formocresol Pulpotomy
  Arms: Pulpotomy using Formocresol

SUMMARY:
The goal of this clinical trial is to evaluate whether Chitosan liquid will show similar clinical and radiographical success rate compared to Formocresol when used in vital pulp therapy in primary molars.

The main question it aims to answer is:

* Will Chitosan liquid, in comparison to Formocresol, show similar clinical outcomes in relation to presence/absence of post-operative pain, swelling, sinus and/or fistula formation when used in vital pulpotomy in primary molars?
* Will Chitosan liquid, in comparison to Formocresol, show similar radiographical outcomes in relation to presence/absence of furcal involvement, periapical lesion, pathological root resorption and/or widening of periodontal membrane space when used in vital pulpotomy in primary molars?

Following conventional pulpotomy procedure, the primary investigator will evaluate the effect of placing a cotton pellet damp with Chitosan liquid directly on radicular vital pulp compared to that of placing a cotton pellet damp with Formocresol on radicular vital pulp.

Primary teeth included in both arms of the study will be restored by zinc oxide and eugenol and covered by a stainless steel crown as final restoration.

The clinical trail will be followed up for 1 year. Clinical outcomes will be evaluated every 3 months. Radiographic outcomes will be evaluated every 6 months.

DETAILED DESCRIPTION:
The main goal of pulp therapy is to maintain the integrity and health of the teeth and their supporting tissues while ensuring the vitality of the pulp of a tooth affected by caries, traumatic injury, or other causes.

Formocresol is a favored medicament for pulp therapy due to its proven success as a fixative, disinfectant, and devitalizing agent. For the past 70 years, it has been the most popular agent for vital pulpotomy in deciduous teeth with a success rate between 70-98%. However, concerns were issued about the potential toxic, mutagenic and cytotoxic effects of formocresol use.

Chitosan is a polysaccharide obtained by alkaline de-acetylation of chitin which is a very common natural biopolymer that can be found in the exoskeleton of crustacea. Chitosan is extensively studied in medical and pharmaceutical fields due to its competitive biological properties like biocompatibility, nontoxicity, analgesic, antitumor, hemostatic, antimicrobial, and antioxidant effects that makes it very interesting to develop for application in dentistry

The aim of the study is to evaluate the clinical and radiographical efficacy of chitosan liquid as pulp medicament compared to formocresol in vital pulpotomy of lower deciduous molars.

In this clinical trial, the principal investigator will carry out all treatment procedures, and the patients will be randomly assigned to any of the intervention groups. For both interventions, informed consent will be obtained from parents/guardians of the participating children.

For both interventions (1 experimental arm group and 1 active comparator arm group):

* Diagnosis of the cases will be performed according to guidelines by the American Academy of Pediatric Dentistry for treatment of vital pulp therapy in primary teeth and a diagnostic chart with personal, medical and dental history will be filled.
* Clinical examination will be done in the dental clinic using mirror and probe to assess the clinical inclusion criteria.
* Preoperative periapical radiographs will be taken to assess the inclusion criteria. Preoperative radiograph will serve as a reference for the follow-up radiographs.
* Baseline records (personal data collection, photographs, percussion test and preoperative periapical radiographs) will be taken.
* An individual Extension Cone Paralleling index will be prepared for each patient by registering the bite through alginate impression and fabricating an acrylic radiographic stent from the patient's cast to allow consistent comparisons of the radiographs.
* Before starting intra-operative procedures, the tooth is allocated randomly (concealed by withdrawing a sealed opaque envelope containing four-folded numbered papers containing the type of dressing material that will be used then writing the patient's name and I.D. on it and will be opened after performing the access cavity).
* Apply topical anesthesia.
* Local anesthesia administration.
* Rubber dam application and access cavity preparation will be established using a sterile bur.
* The envelope marked by the patient's name and I.D. will be opened and the tooth will be allocated into either one of the groups alternatively depending on the pulpotomy medicament used either into Group I (Experimental group) or Group II (Control group)

Group I (Experimental group) pulpotomy using chitosan liquid:

1. After complete hemostasis, a cotton pellet damp with chitosan liquid will be applied and gently placed over the pulp stumps for 5 minutes and removed. Then, a thick mix of zinc oxide and eugenol will be placed and gently condensed into the pulp chamber by a moistened cotton pellet.
2. Tooth will be restored with stainless steel crown.

Group II (Control group) pulpotomy using formocresol:

1. After complete hemostasis, a cotton pellet damp with formocresol will be applied and gently placed over the pulp stumps for 5 minutes and removed. Then, a thick mix of zinc oxide and eugenol will be placed and gently condensed into the pulp chamber by a moistened cotton pellet.
2. Tooth will be restored with stainless steel crown.

The participants are recalled for clinical evaluation at the interval of 3, 6, 9, 12 months, and recalled for radiographic evaluation at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy cooperative children with at least one deep carious mandibular primary molar indicated for vital pulpotomy.
* In age range from 4 to 8 years old.
* Both sexes will be included.
* Patients with provoked pain.
* Restorable teeth.

Exclusion Criteria:

* Excessive haemorrhage that cannot be stopped by a damp cotton pellet after several minutes.
* With congenital anomalies in teeth e.g., taurodontism, concrescence or fusion.
* Patients who show allergic reaction to any material will be used in this trial.
* Will not be able to stick to follow up protocol in the trial and refuse to give communication data.
* Patient's guardians refuse to sign up an informed consent before participating in this trial.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in regards to post-operative pain (spontaneous or on biting) at 3 months | Baseline and 3 months
  Asking the patient and/or guardian to report any pain history at that time frame and/or complaint of discomfort and pain clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to post-operative pain (spontaneous or on biting) at 6 months | Baseline and 6 months
  Asking the patient and/or guardian to report any pain history at that time frame and/or complaint of discomfort and pain clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to post-operative pain (spontaneous or on biting) at 9 months | Baseline and 9 months
  Asking the patient and/or guardian to report any pain history at that time frame and/or complaint of discomfort and pain clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to post-operative pain (spontaneous or on biting) at 12 months | Baseline and 12 months
  Asking the patient and/or guardian to report any pain history at that time frame and/or complaint of discomfort and pain clinically. Outcome measuring unit: Binary (present/absent)

SECONDARY OUTCOMES:
Change from Baseline in regards to swelling at 3 months | Baseline and 3 months
  Visual examination for any sign of redness or swelling of the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to swelling at 6 months | Baseline and 6 months
  Visual examination for any sign of redness or swelling of the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to swelling at 9 months | Baseline and 9 months
  Visual examination for any sign of redness or swelling of the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to swelling at 12 months | Baseline and 12 months
  Visual examination for any sign of redness or swelling of the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to sinus or fistula at 3 months | Baseline and 3 months
  Visual examination for any sign of a sinus or fistula in the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to sinus or fistula at 6 months | Baseline and 6 months
  Visual examination for any sign of a sinus or fistula in the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to sinus or fistula at 9 months | Baseline and 9 months
  Visual examination for any sign of a sinus or fistula in the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to sinus or fistula at 12 months | Baseline and 12 months
  Visual examination for any sign of a sinus or fistula in the gingiva at that time frame and clinically. Outcome measuring unit: Binary (present/absent)
Change from Baseline in regards to furcal lesion at 6 months using Furcation Involvement Scores | Baseline and 6 months
  Radiographic evaluation by visual interpretation of DIGORA software for any furcal lesion using Furcation Involvement Scores. Possible scores range from 0 (no radiolucency) ; 1 (radiolucency between ¼ of furcation to periapical areas); 2 (radiolucency between ¼ to ½ of furcation to periapical areas); 3 (radiolucency more than ½ of furcation to periapical areas).
Change from Baseline in regards to furcal lesion at 12 months using Furcation Involvement Scores | Baseline and 12 months
  Radiographic evaluation by visual interpretation of DIGORA software for any furcal lesion using Furcation Involvement Scores. Possible scores range from 0 (no radiolucency) ; 1 (radiolucency between ¼ of furcation to periapical areas); 2 (radiolucency between ¼ to ½ of furcation to periapical areas); 3 (radiolucency more than ½ of furcation to periapical areas).
Change from Baseline in regards to periapical lesion at 6 months | Baseline and 6 months
  Radiographic evaluation by visual interpretation of DIGORA software for any periapical lesion, cyst formation or obliteration.
Change from Baseline in regards to periapical lesion at 12 months | Baseline and 12 months
  Radiographic evaluation by visual interpretation of DIGORA software for any periapical lesion, cyst formation or obliteration.
Change from Baseline in regards to pathologic root resorption at 6 months | Baseline and 6 months
  Radiographic evaluation by visual interpretation of DIGORA software for any internal, external, early or pathologic root resorption from periapical radiographs.
Change from Baseline in regards to pathologic root resorption at 12 months | Baseline and 12 months
  Radiographic evaluation by visual interpretation of DIGORA software for any internal, external, early or pathologic root resorption from periapical radiographs.
Change from Baseline in regards to width of periodontal membrane space at 6 months | Baseline and 6 months
  Radiographic evaluation by visual interpretation of DIGORA software for any widening in periodontal membrane space from periapical radiographs.
Change from Baseline in regards to width of periodontal membrane space at 12 months | Baseline and 12 months
  Radiographic evaluation by visual interpretation of DIGORA software for any widening in periodontal membrane space from periapical radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No